CLINICAL TRIAL: NCT04099199
Title: A Healthcare Economic Study of the Click Sexual Health Test
Acronym: HERO
Status: Completed | Type: Observational
Sponsor: Visby Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-000274
Record Dates: First submitted 2019-09-12; First posted 2019-09-23 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Click Sexual Health Test — The Click Diagnostics device is a single-use (disposable), fully integrated, rapid, compact, device containing a polymerase chain reaction (PCR)-based nucleic acid amplification test (NAAT) for accurate, qualitative detection and differentiation of deoxyribonucleic acid (DNA) for Neisseria gonorrhea (NG), Trichomonas vaginalis (TV), and Chlamydia trachomatis (CT) organisms.

SUMMARY:
This is a multicenter study with a minimum of three CLIA-Waived intended operator sites in which prospectively collected vaginal swab specimens will be evaluated with the Click Sexual Health Test as compared to standard of care. The specimen collection will occur over one study visit for each enrolled subject, but study staff will continue to follow the subject through standard of care until the subject receives treatment or she is lost to follow up.

ELIGIBILITY:
Inclusion Criteria:

* Documentation that the subject has provided informed consent prior to conducting study procedures
* Subject is symptomatic or asymptomatic for sexually transmitted infections
* Subject is female and 14 years of age or older at the time of enrollment
* Able and willing to follow study procedures

Exclusion Criteria:

* Subject has been previously enrolled in the study
* Subject has a contraindication, medical condition, serious intercurrent illness or other circumstance that in the investigator's judgement, could jeopordize the subject's safety or could interfere with the study procedures
* Use of antiperspirants and deodorants or the following vaginal products: douches, washes, lubricants, vaginal wipes, vaginal moisturizers, or feminine hygiene spray in the genital area, within 48 hours prior to enrollment.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises female subjects greater than or equal to 14 years of age who may be symptomatic or asymptomatic for sexually transmitted infections at locations including, but not limited to: physician offices, OB/GYN, emergency department, and urgent care. Any subject who meets the eligibility will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Benefits of the Click Device for the detection of CT, NG, and TV in self-collected vaginal specimens as compared to standard of care | up to 1 month
Costs of the Click Device for the detection of CT, NG, and TV in self-collected vaginal specimens as compared to standard of care | up to 1 month
Cost-effectiveness of the Click Device for the detection of CT, NG, and TV in self-collected vaginal specimens as compared to standard of care | up to 1 month
Preferences of the Click Device for the detection of CT, NG, and TV in self-collected vaginal specimens as compared to standard of care | up to 1 month
Usability of the Click Device for the detection of CT, NG, and TV in self-collected vaginal specimens as compared to standard of care | up to 1 month
Accuracy of treatment/no treatment decisions in light of the outcomes of testing for CT, NG, and TV infections by Click device as compared to standard of care | up to 1 month
Usability and Satisfaction will be measured by 5-point Likert scale responses, yes/no questions, and open-text questions from study subjects, study operators, and healthcare providers. | up to 1 month
  The scale measures responses to questions in the form of: (1) Strongly Disagree, (2) Disagree, (3) Neutral, (4) Agree, and (5) Strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Health, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dawkins M, Bishop L, Walker P, Otmaskin D, Ying J, Schmidt R, Harnett G, Abraham T, Gaydos CA, Schoolnik G, DiBenedetto K. Clinical Integration of a Highly Accurate Polymerase Chain Reaction Point-of-Care Test Can Inform Immediate Treatment Decisions for Chlamydia, Gonorrhea, and Trichomonas. Sex Transm Dis. 2022 Apr 1;49(4):262-267. doi: 10.1097/OLQ.0000000000001586. PMID 34813579